CLINICAL TRIAL: NCT02386189
Title: Dual Health Systems Users: Strategies to Implement Optimal Care Coordination
Brief Title: Pilot Study to Improve Care Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SDR 14-392
Record Dates: First submitted 2015-02-11; First posted 2015-03-11 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Illness
Keywords: Continuity of Patient Care; Health Records, Personal; Veterans; Patient Participation; Chronic Disease
MeSH Terms: conditions — Chronic Disease; Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: For one of the outcomes (laboratory duplication) the assessor is blind to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Veterans randomized to usual care will not receive any training on using their patient portal(s) to access and share information. They will be contacted via phone and/or secure messaging to remind him/her to take the VA or non-VA provider packet to their appointment. At the conclusion of the study, Veterans assigned to usual care will be provided the training information on the VA health summary for their own reference.
- Care Coordination (Active Comparator): Veterans in this group will share a comprehensive list of all of their providers (VA and non-VA) at future appointments. He/she will also be trained on how to create a VA Health Summary in My HealtheVet to share with their non-VA providers and how to use their community portals (if available) to share information back to VA providers. A VA and non-VA provider visit will be evaluated.
  Interventions: Behavioral: Patient Care Coordination Training

INTERVENTIONS:
Behavioral: Patient Care Coordination Training — Veterans in this group will share a comprehensive list of all of their providers (VA and non-VA) at future appointments. He/she will also be trained on how to create a VA Health Summary in My HealtheVet to share with their non-VA providers and how to use their community portals (if available) to share information back to VA providers. A VA and non-VA provider visit will be evaluated.
  Arms: Care Coordination

SUMMARY:
The purpose of this study is 1) to learn how VA patients can help share their health information between their VA providers and providers outside the VA and 2) if sharing this information is useful to providers and improves care received.

DETAILED DESCRIPTION:
Recent studies estimate that 43 to 75% of Veterans also receive care from non-VA providers (dual use). Dual use is a concern because splitting care between two or more health systems and multiple providers may result in poor coordination of services and a loss of continuity -ultimately putting the patient at increased risk for poor outcomes. Addressing dual use in Veterans is an issue of care coordination. One component of care coordination is information sharing, which often relies on the patient to share information between systems/providers. Veterans registered in My HealtheVet with premium account status have access to download and print a VA health summary (VA CCD). This health summary can be shared with non-VA providers to inform them about recent VA care. This pilot randomized controlled trial will compare usual care to an intervention which aims to improve care coordination for dual use Veterans by educating them about the use of information technology to share health information and informing their providers about the extent and nature of care from other health care systems.

Methods: Dual use Veterans with at least one chronic health condition and both an upcoming VA and non-VA appointments within the study time frame will be eligible to participate. Veterans will be randomized to the intervention or usual care. Veterans in the intervention group will be trained on use of My HealtheVet and their community patient portal (if applicable) to access summary health information to share with providers. In addition, he/she will create a document that lists all members of their health care team. All participants will be asked to take a provider evaluation packet each provider visit (VA and non-VA). After the visit, a phone call will be scheduled with the Veteran to ask about the appointment and medical records from the appointment will be obtained. Outcomes: The main outcomes will be related to patient perceived continuity of care, provider relational coordination survey, medication concordance, and medical laboratory test duplication. Pre and post scores on the patient activation measures will also be explored.

ELIGIBILITY:
Inclusion Criteria:

VA Patient

* Receives health care from VA and non-VA provider
* Diagnosed with a chronic health condition
* Prescribed 5 or more medications
* Upcoming VA and non-VA appointments within the study time frame
* Registered or willing to become registered with My HealtheVet
* Access to a computer with internet, phone, and a printer.
* English speaking

VA or Non-VA Providers: provide care to a stuy participant

Exclusion Criteria:

* Previously shared health data with a provider via their My HealtheVet or local provider patient portal
* No scheduled VA or non-VA appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L Turvey, PhD MS, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haggerty JL, Roberge D, Freeman GK, Beaulieu C, Breton M. Validation of a generic measure of continuity of care: when patients encounter several clinicians. Ann Fam Med. 2012 Sep-Oct;10(5):443-51. doi: 10.1370/afm.1378. PMID 22966108
- [Background] Manski-Nankervis JA, Blackberry I, Young D, O'Neal D, Patterson E, Furler J. Relational coordination amongst health professionals involved in insulin initiation for people with type 2 diabetes in general practice: an exploratory survey. BMC Health Serv Res. 2014 Nov 1;14:515. doi: 10.1186/s12913-014-0515-3. PMID 25361788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects, identified through VA administrative data, were recruited by mail.
Period: Overall Study
Arm/Group | Usual Care | Care Coordination
Started | 30 | 33
Completed | 26 | 30
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Veterans who have sought care within the local VA Health Care System
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Care Coordination | Total
Number analyzed (Participants) | 26 | 30 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 22 | 24 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 24 | 27 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 30 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 25 | 30 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 30 | 56

OUTCOME MEASURES:

1. Primary Outcome: Patient Perceived Continuity of Care From Multiple Providers- Management Continuity
Description: Patient Perceived Continuity of Care was assessed using Haggerty's measure of the same title. Management continuity refers to the patient being able to identify one provider who is the main coordinator and assures all the links within the health care team. The possible range on this measure was between 5 and 40 and the analysis was conducted on the pre-post difference on Management Continuity, subtracting the baseline score from the post-intervention score. More positive score indicated greater perceived management continuity and greater improvement in perceived management continuity.
Time Frame: The time frame is from baseline assessment to 12 months post baseline during which at least one VA and one Community medical visit occurred.
Population: All participants who completed the study and had both a baseline and 12-month follow-up assessment of Patient Perceived Continuity of Care from Multiple Providers. A positive score indicates improvement on this measure over the study period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Care Coordination
Number analyzed (Participants) | 26 | 28
units on a scale | -0.65 (6.4) | 4.0 (8.1)
Statistical Analysis 1: Comparison: Usual Care vs Care Coordination; The t-test was conducted on change between baseline and 12-month follow-up; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Net) = -4.65, Standard Deviation 7.3

2. Primary Outcome: Patient Perceived Continuity of Care From Multiple Clinicians - Informational Continuity
Description: Patient Perceived Continuity of Care was assessed using Haggerty's measure of the same title. Informational Continuity refers to whether patients experienced communication failures between providers. The possible range on this measure was between 12 and 36. The analysis was conducted on the pre-post difference on Informational Continuity, subtracting the baseline score from the post-intervention score. For this measure a lower score and a decline between post intervention and baseline scores (or a negative value) indicates more positive outcomes.
Time Frame: Baseline to 12-month follow-up
Population: All study participants with a baseline and 12-month follow-up assessment completed of Haggerty's Patient Perceived Continuity of Care from Multiple Clinicians.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Care Coordination
Number analyzed (Participants) | 26 | 28
units on a scale | 2.3 (5.6) | -0.59 (5.3)
Statistical Analysis 1: Comparison: Usual Care vs Care Coordination; Test type: Superiority; p = 0.06, t-test, 2 sided; Mean Difference (Net) = 2.91, Standard Deviation 5.5

3. Primary Outcome: Patient Perceived Continuity of Care From Multiple Clinicians- Role Continuity
Description: Patient Perceived Continuity of Care was assessed using Haggerty's measure of the same title. Role Continuity refers to the role of all clinicians being clear to the patient and to the providers on the treatment team. The possible range on this measure was between 6 and 30, and the analysis was conducted on the pre-post difference on this measure. More positive score indicated greater perceived role clarity and, when comparing pre and post score, a more positive score indicated greater improvement in perceived role clarity.
Time Frame: Baseline to 12-month follow-up
Population: All participants who had a baseline and 12- month follow-up assessment of the Patient Perceived Continuity of Care from Multiple Clinicians.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Care Coordination
Number analyzed (Participants) | 26 | 28
units on a scale | -0.04 (2.7) | -0.32 (2.8)
Statistical Analysis 1: Comparison: Usual Care vs Care Coordination; Test type: Superiority; p = 0.71, t-test, 2 sided; Mean Difference (Net) = 0.28, Standard Deviation 2.7

4. Secondary Outcome: Number of Participants With Duplication of Laboratory Tests
Description: Participants had at least one VA medical visit and one community medical visit. Medical records were obtained from both visits and compared. Patients were considered to have a laboratory duplication if the same labs were drawn at both visits and the two visits occurred within three months of each other.
Time Frame: Baseline assessment to 12 months post-baseline, where a laboratory duplication is only counted if the medical visits occurred within three months of each other.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Care Coordination
Number analyzed (Participants) | 26 | 30
Participants | 4 | 1
Statistical Analysis 1: Comparison: Usual Care vs Care Coordination; Test type: Superiority; p = 0.17, Fisher Exact

5. Secondary Outcome: Proportion of Medication Concordance
Description: All participants had at least one VA medical visit and one community medical visit. Medical records were obtained from both visits. Medication lists were obtained from both visits. A medication concordance metric (proportion) was calculated where the denominator was the total number of unique medications identified on both the VA medication list and the community provider medication list. The numerator was the total number of medications (including dose and frequency) that were concordant between the medication lists. This comparison did not include over the counter medications.
Time Frame: Time frame between two medical visits occuring within the one year study period
Population: This sample is based on all participants for whom we had both the VA medication list and the community provider list. We obtained the VA medication list for all, but did not receive all medical records from community providers even after repeated requests.
Measure: Mean (Standard Deviation); unit: Proportion of medications concordant
Arm/Group | Usual Care | Care Coordination
Number analyzed (Participants) | 25 | 30
Proportion of medications concordant | 0.33 (0.15) | 0.34 (0.14)
Statistical Analysis 1: Comparison: Usual Care vs Care Coordination; Test type: Superiority; p = 0.75, t-test, 2 sided; Mean Difference (Net) = -0.01, Standard Deviation 0.15

6. Secondary Outcome: Relational Coordination- VA Providers
Description: Relational Coordination was assessed using Gittell's 7-item measure as described Relational coordination amongst health professionals involved in insulin initiation for people with type 2 diabetes in general practice: an exploratory survey. This was assessed by providers seeing patients enrolled in this study, and this outcome is based on VA providers assessment of Relational Coordination. The scale total score could range from 7 to 35 with higher scores indicating greater relational coordination.
Time Frame: Providers completed the coordination measure at the time of the medical visit which could occur at any point in the 12 month follow-up period.
Population: Veterans gave providers this measure at the medical visit and asked them to complete it and mail it to the study team.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Care Coordination
Number analyzed (Participants) | 15 | 14
units on a scale | 14.9 (6.8) | 18.6 (7.3)
Statistical Analysis 1: Comparison: Usual Care vs Care Coordination; Test type: Superiority; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = -3.6, Standard Deviation 7.1

7. Secondary Outcome: Relational Coordination Community Providers
Description: Relational Coordination was assessed using Gittell's 7-item measure as described iRelational coordination amongst health professionals involved in insulin initiation for people with type 2 diabetes in general practice: an exploratory survey. The scale total score could range from 7 to 35 with higher scores indicating greater relational coordination.
Time Frame: as for outcome 6
Population: This analysis population is based on community providers who actually returned the assessment provided by the patient.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Care Coordination
Number analyzed (Participants) | 10 | 16
units on a scale | 13.5 (9.2) | 14.0 (8.9)
Statistical Analysis 1: Comparison: Usual Care vs Care Coordination; Test type: Superiority; p = 0.89, t-test, 2 sided; Mean Difference (Final Values) = -0.5, Standard Deviation 8.9

ADVERSE EVENTS:
Time Frame: 12 month period
Arm/Group | Usual Care | Care Coordination
All-Cause Mortality (participants affected / at risk) | 1/26 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/30
Other Adverse Events (participants affected / at risk) | 0/26 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=26) | Care Coordination (N=30)
death (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The main limitation is that this is a pilot study and thus has a small sample size.

Another limitation is the poor response rate from providers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT02386189/Prot_SAP_000.pdf